CLINICAL TRIAL: NCT04379401
Title: Acute Impact of Cardiac Resynchronization on Vascular Function (RVA-CRT)
Acronym: RVA-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andreas Flammer (Other)
Responsible Party: Sponsor-Investigator, Andreas Flammer, PD Dr. med. Andreas Flammer, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: RVACRT
Record Dates: First submitted 2020-01-30; First posted 2020-05-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Intervention Model Description: Clinical study with a randomized (double-blind) cross-over design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biventricular Pacing deactivated (Other): The primary objective of the study is to determine, whether short term activation/deactivation of biventricular pacing (BivP) of the CRT (during routine CRT interrogation) has an effect on vascular function
  Interventions: Device: Cardiac Resynchronization Therapy (ON vs. OFF)
- Biventricular Pacing activated (Other): The primary objective of the study is to determine, whether short term activation/deactivation of biventricular pacing (BivP) of the CRT (during routine CRT interrogation) has an effect on vascular function
  Interventions: Device: Cardiac Resynchronization Therapy (ON vs. OFF)

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy (ON vs. OFF) — This study involves study participants, who already received cardiac resynchronisation therapy implantation for clinical reasons. CRT is authorized for medical use by Swissmedic in Switzerland and all implanted devices are CE-approved.

SUMMARY:
Evaluation of the effect of short term activation/deactivation of biventricular pacing (BivP) of the CRT (during routine CRT interrogation) on vascular function as assessed via retinal vessel analysis (RVA), in patients treated with CRT.

DETAILED DESCRIPTION:
Heart failure is a condition in which the heart becomes unable to maintain the body's need of blood supply. Congestive heart failure can be considered a syndrome but the final common path of many cardiovascular diseases. Recently, the investigators of this study confirmed an increased impairment in retinal microvascular function in patients with ischemic heart failure compared to patients with stable coronary disease.

If medication fails to improve ejection fraction, cardiac resynchronization therapy (CRT) is the guideline-recommended treatment for patients with advanced heart failure and bundle branch block.

The question remains if CRT changes purely hemodynamics by synchronizing the heart or has potential impact on the microvasculature to cause reverse remodeling of the failing heart. Measuring retinal vascular function might increase knowledge on the effects of cardiac resynchronization therapy.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Patients ≥ 18 years of age, male or female, diagnosed with advanced heart failure
* Implanted as well as activated CRT device for at least 3 months prior to Visit 1

Exclusion Criteria:

* Current acute decompensated HF
* Documented pacing dependency
* Documented AV-Block II (Mobitz Typ 2) or III in patient's history
* History of hypersensitivity or allergy to Tropicamide
* Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or other major cardiovascular (CV) surgery, percutaneous coronary intervention (PCI) or carotid angioplasty within 3 months prior to Visit 1.
* History of heart transplant, on a transplant list or with ventricular assistance device (VAD).
* Presence of any other disease with a life expectancy of < 6 months
* Presence of significant endocrine diseases, including primary hyperparathyroidism, Cushing's disease, adrenal insufficiency, pituitary tumors, primary hyperaldosteronism, manifest hyperthyroidism or genetic endocrine disorders
* Presence of active acute infectious diseases.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc
* Women who are pregnant or breast feeding
* Known narrow-angle glaucoma
* Known epilepsy (flicker-light could trigger a seizure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Flicker-light induced vasodilatation of retinal arterioles assessed by retinal vessel analyzer (RVA) | A single study 1 day visit is planned.
  Difference in flicker-light induced vasodilatation of retinal arterioles between biventricular pacing of the CRT switched ON and OFF.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas J Flammer, MD, Principal Investigator — University of Zurich
Locations (1):
- UniversitätsSpital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet decided in what way there will be data sharing.